CLINICAL TRIAL: NCT02332655
Title: Cannabidiol Expanded Access Study in Medically Refractory Sturge-Weber Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Anne Comi, MD (Other)
Collaborators: Jazz Pharmaceuticals (Industry); Faneca 66 Foundation (Other)
Responsible Party: Sponsor-Investigator, Anne Comi, MD, Principal Investigator, Director Sturge-Weber Center, Kennedy Krieger Institute, Professor Johns Hopkins University School of Medicine, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Organization: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00029264
Record Dates: First submitted 2015-01-05; First posted 2015-01-07 (Estimated); Results first posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Sturge-Weber Syndrome
Keywords: Sturge-Weber syndrome; SWS; Drug resistant epilepsy
MeSH Terms: conditions — Sturge-Weber Syndrome; Drug Resistant Epilepsy | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cannabidiol (Experimental): All subjects will receive the experimental Epidiolex (cannabidiol) oral solution to be taken at home twice a day, and will be treated on an outpatient basis. The drug will be taken for 48 weeks unless the subject chooses to participate in the extension phase of the study, in which case the subject will continue to receive the drug for one additional year or until the drug is approved for clinical use for the treatment of epilepsy in patients with Sturge-Weber syndrome.
  Interventions: Drug: Cannabidiol

INTERVENTIONS:
Drug: Cannabidiol — Initiation of treatment will begin with 2mg/kg/day. The dose will be increased by 3 mg/kg/day after seven days and then by 5 mg/kg/day every seven days up to a maximum dose of 25 mg/kg/day given.
  The dose of concomitant antiepileptic drugs will remain unchanged during the first 12 weeks of CBD treatment (or until 8 weeks after steady state at final dose), unless symptoms of toxicity and/or significant changes in blood levels are observed.
  Other Names: Epidiolex; CBD

SUMMARY:
The purpose of this study is to determine the tolerability and optimal dose of cannabidiol (CBD) as an simultaneous treatment in children and young adults with Sturge-Weber syndrome (SWS) and drug resistant epilepsy.

DETAILED DESCRIPTION:
We hope to gain an understanding of the utility of pure CBD used for the treatment of medically refractory epilepsy in SWS in this open-label, safety dose-finding, study. Recent evidence suggests that CBD has multiple, beneficial, effects in patients (such as those with SWS that undergo neurological deterioration) suffering from medically refractory seizures. We hypothesize that CBD will reduce seizure frequency in children and young adults with SWS and will therefore help stabilize and improve their neurologic status.This trial is part of an expanded access program, available through a partnership with GW Pharmaceutical, which has been sanctioned by the FDA to study the safety and efficacy of Epidiolex (cannabidiol/CBD) in participants with SWS and medically refractory seizures.

ELIGIBILITY:
Inclusion Criteria: Participants with Sturge-Weber syndrome brain involvement as defined on neuroimaging (n=10 subjects, male and female, ages 1 month to 45 years of age) and the following:

* Documentation of a diagnosis of drug resistant epilepsy as evidenced by failure to control seizures despite appropriate trial of two or more AEDs at therapeutic doses. Drug resistant epilepsy for this study is defined as: At least 1 reported quantifiable (no cluster or innumerable) defined seizure with motor signs per month for at least 3 months prior to initial visit and during the period between Visit 1 (Screening Visit) and Visit 2 (Baseline Visit), as per data captured in daily seizure diaries. These can be focal seizures, focal seizures with impaired consciousness, myoclonic seizures, generalized, and secondarily generalized seizures.
* Between 1-5 baseline anti-epileptic drugs at stable doses for a minimum of 4 weeks prior to enrollment. Vagus nerve stimulator (VNS), ketogenic diet and modified Atkins diet do not count toward this limit.
* VNS must be on stable settings for a minimum of 3 months prior to enrollment.
* If on ketogenic or Atkins diet, must be on stable ratio for a minimum of 3 months prior to enrollment.
* Previous subjects who failed at any point to meet continuation criteria and withdrew early may be considered for re-enrollment under a new subject ID as long as the above inclusion criteria are met. The determination of whether to re-enroll will be made by the PI and sponsor on a case-by-case basis. Re-enrollment can occur no earlier than 4 weeks after the final, post-weaning follow-up visit under the old subject ID.

Written informed consent obtained from the patient or the patient's legal representative must be obtained prior to beginning treatment.

Exclusion Criteria:

* Patients with seizures secondary to metabolic, toxic, infectious or psychogenic disorder or drug abuse or current seizures related to an acute medical illness.
* Presence of only non-motor partial seizures (without limb or facial movements, eye deviation or head turning)
* Patients who require rescue medication during the Baseline phase for more than 6 days.
* Patients with any severe and/or uncontrolled medical conditions at randomization such as:

  1. liver disease such as cirrhosis, decompensated liver disease, and chronic hepatitis [i.e. quantifiable hepatitis B virus (HBV)-DNA and/or positive HbsAg, quantifiable hepatitis C virus (HCV)-RNA]
  2. Uncontrolled diabetes as defined by fasting serum glucose > 1.5
  3. Active (acute or chronic) or uncontrolled severe infections.
  4. Patients with an active, bleeding diathesis.
* Patients who have had a major surgery or significant traumatic injury within 4 weeks of study entry. Patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia), or patients that may require major surgery during the course of the study.
* Patients who change the dose of the AEDs during 4 weeks before screening or during the baseline period.
* Prior treatment with any investigational drug within the preceding 4 weeks prior to study entry.
* Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will not be able to complete the entire study. Those in foster care, unable to keep follow-up appointments, maintain close contact with Principal Investigator, or complete all necessary studies to maintain safety.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test.

Ages: 1 Month to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2014-12; Primary Completion 2019-04 (Actual); Study Completion 2021-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne M Comi, MD, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

REFERENCES:
- See also: Hunter Nelson Sturge-Weber Center Website — http://www.kennedykrieger.org/patient-care/patient-care-centers/sturge-weber-center

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All enrolled participants will receive cannabidiol.
Groups:
- Cannabidiol: All subjects will receive the experimental Epidiolex (cannabidiol) oral solution to be taken at home twice a day, and will be treated on an outpatient basis. The drug will be taken for 48 weeks unless the subject chooses to participate in the extension phase of the study, in which case the subject will continue to receive the drug for one additional year or until the drug is approved for clinical use for the treatment of epilepsy in patients with Sturge-Weber syndrome.
  Cannabidiol: Initiation of treatment will begin with 2mg/kg/day. The dose will be increased by 3 mg/kg/day after seven days and then by 5 mg/kg/day every seven days up to a maximum dose of 25 mg/kg/day given.
  The dose of concomitant antiepileptic drugs will remain unchanged during the first 12 weeks of CBD treatment (or until 8 weeks after steady state at final dose), unless symptoms of toxicity and/or significant changes in blood levels are observed.
Period: Overall Study
Arm/Group | Cannabidiol
Started | 5
Completed | 4
Not Completed | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cannabidiol
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.83 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Seizures Per Month
Description: A baseline seizure frequency was recorded for each subject in a diary for eight weeks prior to investigational drug initiation and parents/caregivers documented seizures on a daily basis throughout the trial using a seizure log. For assessing the efficacy of CBD, the investigator counted the change in frequency of seizures per month. The number of seizures within 56 days of the baseline and the number of seizures within 56 days of week 14 were calculated. Higher seizure frequency indicates worse outcome. This outcome is measured as the change in number of seizures per month between the baseline and week 14 time points.
Time Frame: Measured within 56 days before baseline and 56 days before week 14
Population: 4 out of 5 subjects were included in analysis as subject 5 was removed early (before week 14) due to lack of efficacy and adverse events.
Measure: Mean (Standard Deviation); unit: Seizures per month
Arm/Group | Cannabidiol
Number analyzed (Participants) | 4
Seizures per month
  Subject 1 Overall Average Number of Seizures per Month at Baseline: number analyzed (Participants) | 1
  Subject 1 Overall Average Number of Seizures per Month at Baseline | 33.5 (7.78)
  Subject 1 Overall Average Number of Seizures per Month at Week 14: number analyzed (Participants) | 1
  Subject 1 Overall Average Number of Seizures per Month at Week 14 | 30.0 (2.83)
  Subject 2 Overall Average Number of Seizures per Month at Baseline: number analyzed (Participants) | 1
  Subject 2 Overall Average Number of Seizures per Month at Baseline | 3.0 (1.41)
  Subject 2 Overall Average Number of Seizures per Month at Week 14: number analyzed (Participants) | 1
  Subject 2 Overall Average Number of Seizures per Month at Week 14 | 0.5 (0.71)
  Subject 3 (Re-enrolled) Overall Average Number of Seizures per Month at Baseline: number analyzed (Participants) | 1
  Subject 3 (Re-enrolled) Overall Average Number of Seizures per Month at Baseline | 3.0 (1.41)
  Subject 3 (Re-enrolled) Overall Average Number of Seizures per Month at Week 14: number analyzed (Participants) | 1
  Subject 3 (Re-enrolled) Overall Average Number of Seizures per Month at Week 14 | 2.0 (0.00)
  Subject 4 Overall Average Number of Seizures per Month at Baseline: number analyzed (Participants) | 1
  Subject 4 Overall Average Number of Seizures per Month at Baseline | 5.0 (1.41)
  Subject 4 Overall Average Number of Seizures per Month at Week 14: number analyzed (Participants) | 1
  Subject 4 Overall Average Number of Seizures per Month at Week 14 | 0.5 (0.71)
  Subject 5 Overall Average Number of Seizures per Month at Baseline: number analyzed (Participants) | 1
  Subject 5 Overall Average Number of Seizures per Month at Baseline | 1.0 (0.00)
  Subject 5 Overall Average Number of Seizures per Month at Week 14: number analyzed (Participants) | 0

2. Secondary Outcome: Percentage Change in Seizure Frequency at Most Recent Visit on CBD Compared With Baseline
Description: The percentage change, between the seizure frequency per month reported at baseline compared to seizure frequency per month at the subject's most recent visit, on CBD was calculated. Higher positive percentage change in seizure frequency per month would indicate better outcome. Positive values indicate a decrease in seizure frequency.
Time Frame: Measured at Baseline and most recent visit within 1 year
Population: 4 out of 5 subjects were included in analysis as subject 5 was removed early due to lack of efficacy. Data were not collected for Subject 5 as the subject was removed at week 9 due to lack of efficacy.
Measure: Number; unit: Percentage Change in Seizure Frequency
Arm/Group | Cannabidiol
Number analyzed (Participants) | 4
Percentage Change in Seizure Frequency
  Subject 1 Percent decrease in Seizure Frequency at Most Recent Visit on CBD Compared with Baseline: number analyzed (Participants) | 1
  Subject 1 Percent decrease in Seizure Frequency at Most Recent Visit on CBD Compared with Baseline | 12
  Subject 2 Percent decrease in Seizure Frequency at Most Recent Visit on CBD Compared with Baseline: number analyzed (Participants) | 1
  Subject 2 Percent decrease in Seizure Frequency at Most Recent Visit on CBD Compared with Baseline | 100
  Subject 3 Percent decrease in Seizure Frequency at Most Recent Visit on CBD Compared with Baseline: number analyzed (Participants) | 1
  Subject 3 Percent decrease in Seizure Frequency at Most Recent Visit on CBD Compared with Baseline | 83
  Subject 4 Percent decrease in Seizure Frequency at Most Recent Visit on CBD Compared with Baseline: number analyzed (Participants) | 1
  Subject 4 Percent decrease in Seizure Frequency at Most Recent Visit on CBD Compared with Baseline | 64
  Subject 5 Percent decrease in Seizure Frequency at Most Recent Visit on CBD Compared with Baseline: number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 48 weeks
Description: All adverse events, unanticipated problems, protocol deviations or other concerns will be promptly reported to the principal or co-investigator who will have primary responsibility for notifying the IRB and the KKI Office of Research Compliance. As stated previously, no serious risks are anticipated. All side effects or adverse events problems of a medical nature will also be reported to GW Pharmaceutical.
Arm/Group | Cannabidiol
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 3/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cannabidiol (N=5)
Left Eye Vertical Nystagmus (Eye disorders) | 1 (1) — Subject reported vertical eye movement in left eye that persisted for several months. Pressures were same as baseline and no change in apparent vision or visual field cut were detected. MRI was conducted and patient was seen for follow up.
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — The participant got sick with vomiting and diarrhea. He had a seizure and was noted to have a cough and fever. After having two more seizures, he was taken to the ER where an x-ray determined he had pneumonia and dehydration.
Facial Skin Infection (Skin and subcutaneous tissue disorders) | 1 (1) — Subject picked at a facial pimple above her left eye. The area reddened and began to swell. She was taken to the ER and given IV antibiotics.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cannabidiol (N=5)
Temporary increased seizures (Nervous system disorders) | 3 (3)
Behavioral Issues (Psychiatric disorders) | 2 (2)
Increased aspartate aminotransferase liver function test (Investigations) | 1 (1)
Right eye exotropia and redness/intermittent exotropia without redness (Eye disorders) | 1 (1)
Tiredness (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-06): https://cdn.clinicaltrials.gov/large-docs/55/NCT02332655/Prot_SAP_000.pdf